CLINICAL TRIAL: NCT02959398
Title: EVALUATION DE LA TOMOSYNTHESE DANS LA CARACTERISATION ET LA PRISE EN CHARGE DES LESIONS MAMMAIRES : "ETOLE"
Brief Title: Evaluation of Tomosynthesis for Characterization and the Management of Breast Lesions
Acronym: ETOLE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: P120121
Record Dates: First submitted 2016-11-07; First posted 2016-11-09 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Breast Neoplasms; Tomosynthesis; BRCA1 Protein; BRCA2 Protein
MeSH Terms: conditions — Breast Neoplasms; Fanconi Anemia, Complementation Group D1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard mammography (Active Comparator): standard mammography
  Interventions: Device: Standard mammography
- standard mammography and tomosynthesis (Experimental): standard mammography and tomosynthesis
  Interventions: Device: Standard mammography and tomosynthesis

INTERVENTIONS:
Device: Standard mammography — Standard mammography
  Arms: standard mammography
Device: Standard mammography and tomosynthesis — Standard mammography and tomosynthesis
  Arms: standard mammography and tomosynthesis

SUMMARY:
Tomosynthesis is an innovative technique developed in digital mammography for obtaining a sectional image of the breast. Mammography has the main disadvantage of being an imaging projection that creates overlays, which eliminates tomosynthesis.

The objective of this study is to evaluate if the BI-RADS classification obtained by tomosynthesis with synthetic mammography is superior to that obtained by conventional mammography in terms of specificity while not inferior in terms of sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Patient having clinical or breast imaging abnormalities classified as BiRads 3, 4, 5 (Table 1). (5)
* Patient over 18 years old
* Signed informed consent

Exclusion Criteria:

* Patients at high risk of breast cancer, mutations BRCA 1 (BReast CAncer gene 1) or BRCA 2 (BReast CAncer gene 2) carriers, Li Fraumeni, or history of thoracic radiation will be excluded because of their greater sensitivity to ionizing radiation.
* Patient unable to give informed consent for physical, mental, or legal reasons.
* Patient not affiliated with French Social Security Insurance.
* Patient under treatment for breast cancer.
* When mammography is not recommended according to good practice by the French Health Authority (HAS).
* Pregnant patient.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2017-11-20 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Breast Imaging-Reporting And Data System (BI-RADS) scale | Day 1
  The primary evaluation parameter will be the classification error of tumors according to the BiRads scale obtained by mammography (BiRadsM) and by tomosynthesis (BiRadsT) according to the gold standard.

SECONDARY OUTCOMES:
Criteria for a poor prognosis | Day 1
  The visibility (presence or absence) of signs of poor prognosis criteria. We will compare the visibility of poor prognosis criteria seen on mammography + ultrasound and seen on tomosynthesis with synthetic mammography + ultrasound.
Number of additional examinations | Day 30
  Needs for supplementary breast imaging exams and biopsies
The number of ultrasound exams | Day 30
Total radiation dose | Day 30
Cost of the diagnostic strategies | Day 30
Agreement between readers | Day 1
  The reproducibility of the interpretation of tomosynthesis will be assessed with differences of classifications BiRadsT observed between the two radiologists
Cumulative incidence of Breast cancer diagnosis | Month 24
  Cumulative incidence of Breast cancer diagnosis among women with benign at after primary evaluation

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - hopital Saint-Louis, Paris
  - Hopital Tenon, Paris